CLINICAL TRIAL: NCT04086342
Title: CHI-902 for Treatment of Social Anxiety Disorder - A Phase IIb Randomized Double-Blind Placebo-Controlled Clinical Trial
Brief Title: CHI-902 for Treatment of Social Anxiety Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes in pipeline
Sponsor: Canopy Growth Corporation (Industry)
Collaborators: Centre for Addiction and Mental Health (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H2017-04
Record Dates: First submitted 2019-08-29; First posted 2019-09-11 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2019-08

CONDITIONS: Social Anxiety Disorder
Keywords: Anxiety; Cannabis; Cannabidiol; CBD
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHI-902 (Active Comparator): Study subjects will enter a titration phase of 1 week with a daily oral CBD dose of 150 mg (50 mg three times daily). Then, daily CBD dose of 300 mg or matching placebo will be given for 3 weeks (treatment phase 1; fixed dose).
  Interventions: Drug: CHI-902
- Placebo (Placebo Comparator): Study subjects will enter a titration phase of 1 week with a daily oral dose of 150 mg (50 mg three times daily) of matching placebo. Then, daily dose of 300 mg of matching placebo will be given for 3 weeks (treatment phase 1; fixed dose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHI-902 — A standardized cannabis extract in MCT oil administered in oral liquid (oil) form.
  Other Names: CBD Oil
  Arms: CHI-902
Drug: Placebo — Placebo is a vehicle oil that will match CHI-902.
  Other Names: Placebo Oil
  Arms: Placebo

SUMMARY:
No substantial clinical trials of Cannabidiol (CBD) in Social Anxiety Disorder (SAD) have yet been conducted. This randomized doubleblind, placebo-controlled trial of CBD in adults with SAD will evaluate the efficacy, tolerability and safety of CBD oil (CHI-902) in SAD. In addition, the effects of treatment with CHI-902 on the Endocannabinoid System (ECS) will be assessed by evaluating peripheral endocannabinoids (Arachidonoylethanolamide/Anandamide (AEA) and 2-Arachidonoyl glycerol (2-AG)) before and after treatment.

DETAILED DESCRIPTION:
This study will evaluate efficacy, therapeutic effects, tolerability and safety of CBD oil in adults with SAD through a randomized placebo-controlled study design and will evaluate effects of CHI-902 on peripheral endocannabinoids (AEA and 2-AG). This study will be the first randomized, double-blind placebo-controlled trial conducted with CHI-902 in adults with SAD.

The study is designed to:

* Evaluate the efficacy of CHI-902 versus placebo in adults with SAD.
* Evaluate the tolerability and safety versus placebo of CHI-902 in adults with SAD.
* Explore the effects of CHI-902 versus placebo on different biomarkers in subjects with SAD.

ELIGIBILITY:
Inclusion Criteria: Adult males or females (≥18 years of age) will be enrolled until the required number of n=160 subjects completing all study procedures is met. Individuals will be included if they:

1. Meet DSM-5 criteria for SAD
2. Score >60 on the Liebowitz Social Anxiety Scale (LSAS)

Exclusion Criteria:

1. Serious, unstable medical condition including but not limited to cerebrovascular, renal, hepatic, coronary heart disease, coagulation/blood disorders, use of anticoagulant medication, pre-existing cardiovascular disease including poorly controlled hypertension, ischaemic heart disease, arrhythmia, or heart failure;
2. Past or current neurological illness or head trauma;
3. History of bipolar disorder, psychotic disorder/schizophrenia, schizoaffective disorder, obsessive-compulsive disorder, or personality disorder (Cluster A or B);
4. Current moderate or severe major depressive episode, panic disorder, generalized anxiety disorder, or post-traumatic stress disorder (PTSD). Traits associated with these disorders are permissible but full DSM criteria should not be met;
5. Current psychotic symptoms;
6. Current suicidal ideation or suicide attempt or self-harm behavior in the past year;
7. Current unstable psychiatric condition;
8. Substance use disorder in the past 6 months except nicotine
9. Cannabis use or use of medications or drugs targeting endocannabinoid system including but not limited to nabiximols, nabilone, or synthetic cannabinoids in the past 3 months;
10. Regular pharmacological treatment with psychotropic medications except benzodiazepines which may be used as a rescue medication
11. Pharmacological treatment with medications with potential significant drug-drug interactions with CBD through Cytochrome P450 metabolization (CYP3A4, CYP2C9, CYP2C19, CYP1A1) based on the Investigator assessment;
12. Pregnancy or lactation;
13. Males and females of child-bearing potential must be using and willing to continue using medically acceptable contraception throughout the study to avoid pregnancy during the study and for up to 4 weeks after study completion, as described below. Study-acceptable methods of birth control are double-barrier methods, which include a combination of any 2 of the following: oral contraceptives, diaphragm, condom, copper intrauterine device, sponge, spermicide, or (partner's) vasectomy;
14. Positive urine during drug screening for drugs of abuse (except benzodiazepines);
15. Reported history of difficulty with intravenous blood draws;
16. Allergy to or intolerability of cannabinoids, CBD or other ingredients of the product;
17. Baseline liver, renal, or hematological laboratory abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-24 (Estimated); Primary Completion 2021-01-26 (Estimated); Study Completion 2021-01-26 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | Baseline to endpoint (week 10)
  Quantitative change in LSAS total score from baseline to endpoint (week 10) in subjects receiving active treatment with CHI-902 compared to subjects receiving placebo.
  The scale is composed of 24 items divided into 2 subscales, 13 concerning performance anxiety, and 11 pertaining to social situations. The 24 items are first rated on a scale from 0 to 3 on fear felt during the situations, and then the same items are rated regarding avoidance of the situation. Combining the total scores for the Fear and Avoidance sections provides an overall score with a maximum of 144 points. Research supports a cut-off point of 30, in which SAD is unlikely. The next cut-off point is at 60, at which SAD is probable. Scores between 60 and 90 indicate that SAD is very probable. Scores higher than 90 indicate that SAD is highly probable.

SECONDARY OUTCOMES:
Systematic Assessment of Side Effects in Clinical Trials (SAFTEE) | After 10 weeks of treatment.
  Safety and adverse effects with the Systematic Assessment for Treatment Emergent Events (SAFTEE). Tolerability of treatment assessed by SAFTEE in subjects receiving active treatment with CHI-902 compared to subjects receiving placebo, and safety through number of subjects dropping out due to SAEs in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ware, MD, Study Director — Canopy Growth Corporation
Locations (2):
- Canada (2):
  - MacAnxiety Research Center, McMaster University, Hamilton, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No